CLINICAL TRIAL: NCT02714465
Title: Treatment of Adverse Radiation Effects After Gamma Knife Radiosurgery (GKS) by Hyperbaric Oxygen Therapy (HBO)
Brief Title: Adverse Radiation Effects After Gamma Knife Radio Surgery and Hyperbaric Oxygen Therapy
Acronym: GKSHBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 644-122015
Record Dates: First submitted 2016-03-01; First posted 2016-03-21 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Necrosis
Keywords: Hyperbaric Oxygen Therapy; Gamma Knife Radiosurgery
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyperbaric oxygen therapy (Experimental): All patients underwent radiosurgery with clinical and instrumental signs of cerebral radionecrosis
  Interventions: Other: hyperbaric oxygen therapy

INTERVENTIONS:
Other: hyperbaric oxygen therapy — hyperbaric oxygen therapy

SUMMARY:
Evaluation of clinical improvement and the reduction of edema lesion documented by magnetic resonance imaging (MRI) in patients with cerebral radiation necrosis post gamma knife surgery (GKS) by treatment with hyperbaric oxygen therapy (HBO)

DETAILED DESCRIPTION:
Patients will be recruited on the basis of the presence of cerebral radionecrosis post gamma knife surgery, documented by both clinical examination (Rankin Scale) and instrumental imaging (MRI). They will be subjected to hyperbaric oxygen therapy HBO, and during treatment the patient performs clinical examination (Rankin Scale) for 24 sessions of HBO. Then they will have a break of 10-15 days during which also performs the instrumental survey (Magnetic Resonance Imaging). If the radionecrosis has regressed they will suspend the treatment otherwise continue up to a maximum of 40 treatment sessions of HBO

ELIGIBILITY:
Inclusion Criteria:

* between 10 and 75 years
* understanding of the Italian language
* ability to understand the procedures and carrying out of the study
* signing informed consent for adults and minors in use
* underwent radiosurgery with clinical and instrumental signs of radiation necrosis

Exclusion Criteria:

* younger than 10yrs old and older than 75yrs old
* not capable to understand Italian language or to understand the protocol procedures and visits' scheme
* informed consent not given
* enrolled in another clinical trial
* concomitant pathologies contraindicate HBO as: emphysema, asthma, epilepsy, claustrophobia; Paul Bert Syndrome, Lorrain Smith Syndrome
* under disulfiram, doxorubicine, cisplatinum, mafenide acetate, bleomycins treatment
* life expectancy less than 6 months
* Rankin Scale >5

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of clinical improvement | day 2 through day 25
  By neurological evaluation (Ranking Scale)

SECONDARY OUTCOMES:
Evaluation of the reduction of the extent of edema lesion documented by MRI | 1-3 months
  MRI analysis
Measurement of complications from hyperbaric oxygen therapy and their severity | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Grande Ospedale Metropolitano Niguarda, Milan, Lombardy, Italy